CLINICAL TRIAL: NCT04934969
Title: The Adjunctive Use of Lavender and Peppermint Essential Oils to Manage Nausea, Pain, and Anxiety in an Adult Orthopedic Population
Brief Title: The Adjunctive Use of Lavender and Peppermint Essential Oils
Acronym: aromatherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Denise Kresevic, clinical nurse specialist, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20190050
Record Dates: First submitted 2021-06-15; First posted 2021-06-22 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Joint Diseases
MeSH Terms: conditions — Joint Diseases | interventions — Aromatherapy

STUDY DESIGN:
Intervention Model Description: feasibility of using essential oils post joint replacement surgery and trends toward relief of symptoms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use of lavender and peppermint essential oils pre and post (Experimental): passive inhalation of either peppermint and lavender essential oil with pre and post test measure
  Interventions: Dietary Supplement: Adjunctive use of lavender and peppermint essential oils

INTERVENTIONS:
Dietary Supplement: Adjunctive use of lavender and peppermint essential oils — passive inhalation aromatherapy following joint surgery
  Other Names: aromatherapy

SUMMARY:
This study will use passive inhalation of lavender for discomfort, anxiety and peppermint for nausea following joint replacement and spine surgery

DETAILED DESCRIPTION:
Following review of records for eligibility and consent obtained during pre op visit subjects will be enrolled in study post op they will validate desire to participate and chose to inhale (2 drops of essential oil on cotton ball in a plastic bag) lavender for discomfort or anxiety or peppermint for GI distress

Visual analogue scales will be used to rate discomfort , anxiety and nausea

ELIGIBILITY:
Inclusion Criteria:

- elective joint replacement able to read and speak English and describe study procedures

Exclusion Criteria:

pregnancy

* unable to smell, sensitivity to fragrances asthma or breathing problems have smoke or vaped in last 2 weeks if atrial fibrillation history no peppermint uncontrolled hypertension above 160/100 non employees of UH or students of CWRU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
discomfort, anxiety, or GI distress | total of 90 minutes
  visual analog sale

CONTACTS AND LOCATIONS:
Overall Officials: Denise Kresevic, PhD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals of Cleveland, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
hope to publish results